CLINICAL TRIAL: NCT05695183
Title: Functionality of the IV SafeLock Device in Emergency Department Setting
Brief Title: IV SafeLock Device Functionality in Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kara J. Bragg, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 22-012282
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Intravenous Access

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emergency Department Nurses (Experimental): Registered nurses will use the IV SafeLock Device on patients during care in the emergency department.
  Interventions: Device: IV SafeLock

INTERVENTIONS:
Device: IV SafeLock — Designed to prevent patient access to intravenous lines in the hospital setting. The device locks with an institution specific key and protects the hub as well as all tubing access points.

SUMMARY:
The purpose of this research study is to evaluate the functionality of the IV SafeLock in the clinical emergency department setting.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Department nurses who are consenting and willing to perform tasks.
* Their patient population will include stable patients 18 or over, who present through triage, are medically stable, are able to verbally consent and require intravenous access.

Exclusion Criteria:

* Emergency Department nurses who are unwilling to consent to use IV SafeLock on their patient population.
* The patient population will exclude pregnant patients, children, prisoners, patients with dementia, or any member of protected class as specified by IRB.
* The patients must be medically stable and not include patients presenting with acute stroke, acute myocardial infarction, severe sepsis or shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-22 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Functionality of the IV SafeLock | Baseline
  Measured on a likert scale for nurse evaluation of IV SafeLock

CONTACTS AND LOCATIONS:
Overall Officials: Kara Bragg, APRN, DNP, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bragg K, Albus M, Bragg B, Beste RM, Simon LV. Evaluation of the Functionality in an Emergency Department Setting of an Intravenous Protection Device to Prevent Self-Injection. Med Devices (Auckl). 2024 Mar 19;17:135-142. doi: 10.2147/MDER.S451439. eCollection 2024. PMID 38529519
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials